CLINICAL TRIAL: NCT07400042
Title: Reducing the Length of Stay and Incidence of Rehospitalization in Heart Failure Patients by Measuring Peripheral Venous Pressure; a Randomized Clinical Trial
Brief Title: Peripheral Venous Pressure (PVP) Randomized Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00142526
Record Dates: First submitted 2026-01-21; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-12

CONDITIONS: Congestive Heart Failure
Keywords: peripheral venous pressure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- peripheral venous pressure measurements (Experimental): Peripheral venous pressure measures provided to physicians daily up to 8 days
  Interventions: Other: peripheral venous pressure measurements
- standard clinical care (Active Comparator): Usual standard clinical care, peripheral venous pressure measures not provided to physician daily
  Interventions: Other: standard clinical care

INTERVENTIONS:
Other: peripheral venous pressure measurements — Peripheral venous pressure measures provided to physicians daily up to 8 days, with a research note in the electronic medical record containing standardized recommendations for case also provided daily. Care changes up to clinical provider discretion.
  Arms: peripheral venous pressure measurements
Other: standard clinical care — Usual standard clinical care
  Arms: standard clinical care

SUMMARY:
The purpose of the study is to determine if there is a reduction in the length of stay and rates of rehospitalization for patients diagnosed with congestive heart failure when physicians are provided daily measurements of peripheral venous pressure versus no daily measurements of peripheral venous pressure.

DETAILED DESCRIPTION:
The objective of the study is to evaluate the effectiveness of standard clinical care versus standard clinical care directed by peripheral venous pressure on length of hospital stay and incidence of rehospitalization among heart failure patients.

The study team hypothesizes that compared to standard clinical care the peripheral venous pressure-guided therapy is associated with shorter hospital stay and lesser incidence of 30-day rehospitalization. The study team will also collect data to determine if peripheral venous pressure-guided care is associated with reduced incidence of 6-month rehospitalization, improvement in symptoms or lab indices, lesser new incidence of dialysis, change in use of diuretics, and lesser use of echocardiograms.

ELIGIBILITY:
Inclusion Criteria:

* Patients with minimum 3-month history of Congestive Heart Failure admitted to Aurora St. Luke's Medical Center with acute decompensation
* English speaking only

Exclusion Criteria:

* Patients who do not already have a peripheral IV line inserted
* Patients whose IV line cannot be transduced
* Patients with current or past vein thrombosis in the arm used to measure the pressure or with history of recurrent (>1) pulmonary embolism
* Patients with active thrombophlebitis in the arm
* Patients who have experienced a major cardiovascular event (myocardial infarction, stroke, etc.) ≤2 months prior to the admission date
* Patients who have received an implanted cardiac resynchronization device (pacemaker or ICD) ≤3 months prior to admission date
* Patients enrolled in other cardiovascular research studies.
* Patients with a clinical condition that the investigator believes may not allow the patient to complete the study, at the discretion of the investigator. Examples of conditions that may apply include severe stenotic valvular disease, isolated right ventricle failure, precapillary pulmonary hypertension, hypertrophic obstructive cardiomyopathy, implanted left ventricular assist device, history of heart transplantation, clinical diagnosis of cardiogenic shock, any left-to-right shunt
* Patients with congenital heart disease or mechanical right heart valve(s)
* Planned heart surgery and/or coronary intervention during hospitalization
* Patients expected to receive heart transplant within 6 months of admission
* IV cannula smaller than 22G
* Patients who are pregnant and/or lactating
* Patients who are unable to provide informed consent
* Patients who are intubated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2041-08 (Estimated); Study Completion 2041-08 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | up to day 8
  Number of days from admission to discharge
Number of subjects rehospitalized | Day 30 post index hospitalization
  Number of subjects in each group who have been rehospitalized
Number of subjects rehospitalized | Month 6 post index hospitalization
  Number of subjects in each group who have been rehospitalized

SECONDARY OUTCOMES:
Number of subjects with exertional dyspnea | Day 1 and date of discharge (up to day 8)
  Number of subjects in each group experiencing dyspnea according to the New York Heart Association Class
Number of subjects with exertional orthopnea | Day 1 and date of discharge (up to day 8)
  Number of subjects in each group experiencing orthopnea according to the New York Heart Association Class
Number of subjects with new need for dialysis during index hospitalization | Day 1 and date of discharge (up to day 8)
  Number of subjects in each group with new need for dialysis during index hospitalization
Number of subjects with diuretic use | Day 1 and date of discharge (up to day 8)
  Number of subjects in each group with diuretic use during index hospitalization
Number of subjects with echocardiograms | Day 1 and date of discharge (up to day 8)
  Number of subjects in each group with echocardiograms performed (with results) during index hospitalization
Number of subjects with all-cause death | Month 6 post index hospitalization
  Number of subjects in each group with all-cause death
Number of subjects with cardiac-related death | Month 6 post index hospitalization
  Number of subjects in each group with cardiac-related death

CONTACTS AND LOCATIONS:
Overall Officials: Khawaja Ammar, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Aurora St. Luke's Medical Center, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No